CLINICAL TRIAL: NCT00280462
Title: Choroidal Blood Flow Regulation During Isometric Exercise: Effects of Ca2+-Channel Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-110705
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Ocular Physiology; Regional Blood Flow
Keywords: Nifedipine; Choroidal blood flow; Choroidal autoregulation; Isometric exercise
MeSH Terms: interventions — Nifedipine; Pharmaceutical Preparations; Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Nifedipine
  Interventions: Drug: Nifedipine (drug); Drug: L-Arginin (drug); Drug: Placebo
- 2 (Active Comparator): L-Arginin
  Interventions: Drug: Nifedipine (drug); Drug: L-Arginin (drug); Drug: Placebo
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Nifedipine (drug); Drug: L-Arginin (drug); Drug: Placebo

INTERVENTIONS:
Drug: Nifedipine (drug) — Nifedipine (Adalat®, Bayer, Leverkusen, Germany) dose: 15µg/kg bolus infusion over 5 minutes; 0.2 µg/(kg.min) maintenance dose infusion period 25 minutes
Drug: L-Arginin (drug) — L-Arginin (Clinalfa AG, Läufelfingen, Switzerland) 30% sodium chlorid solution, dose: 1g/min over 30 minutes
Drug: Placebo — Placebo

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. For a long time it had been assumed that the choroid is a strictly passive vascular bed, which shows no autoregulation. However, recently several groups have identified some autoregulatory capacity of the human choroid. In the brain and the retina the mechanism behind autoregulation is most likely linked to changes in transmural pressure. In this model arterioles change their vascular tone depending on the pressure inside the vessel and outside the vessel. In the choroid, several observations argue against a direct involvement of arterioles. In a previous project we were able to identify that the nitric oxide (NO) - system as well as the endothelin system are involved in choroidal blood flow regulation during isometric exercise.

In the present study autoregulation of the choroid during isometric exercise will be investigated and the pressure/flow relationships will be observed in the absence or presence of a calcium antagonist - nifedipine.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy more than 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Choroidal pressure-blood flow relationship | in total 3x 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjäger-Mayrl, M.D., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Schmidl D, Prinz A, Kolodjaschna J, Polska E, Luksch A, Fuchsjager-Mayrl G, Garhofer G, Schmetterer L. Effect of nifedipine on choroidal blood flow regulation during isometric exercise. Invest Ophthalmol Vis Sci. 2012 Jan 25;53(1):374-8. doi: 10.1167/iovs.11-8536. PMID 22199246